CLINICAL TRIAL: NCT01530412
Title: Long Term Evaluation of Activity Levels Post Pulmonary Rehabilitation: 1 Year Follow-up
Brief Title: Long Term Evaluation of Activity Levels Post Pulmonary Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beaumont Hospital (Other)
Responsible Party: Principal Investigator, Professor Richard Costello, Professor of Medicine, Beaumont Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RCT-3-LTE
Record Dates: First submitted 2010-08-18; First posted 2012-02-10 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2012-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Quality of Life; Free-living activity; Exacerbation; Rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): Patients are randomized to the control group and are assessed pre rehabilitation and post rehabilitation after which they proceed to the intervention group.
- Pulmonary Rehabilitation (Experimental): Patients undergo an active seven week pulmonary rehabilitation programme. Assessments occur pre rehabilitation, post rehabilitation, at three months and at one year.
  Interventions: Other: Pulmonary Rehabilitation

INTERVENTIONS:
Other: Pulmonary Rehabilitation — Patients undergo pulmonary rehabilitation for two hours twice a week for seven weeks. The first hour comprises of an individualized exercise programme and the second hour consists of an educational component. Patients are also required to undergo inspiratory muscle training five days a week for thirty minutes and exercise for an additional three days a week for thirty minutes.
  Arms: Pulmonary Rehabilitation

SUMMARY:
Sustained improvement after pulmonary rehabilitation in activity levels as measured by an activity armband.

Pulmonary rehabilitation is utilized to improve exercise capacity, quality of life and prognosis for patients who suffer from chronic obstructive pulmonary disease. There is also strong evidence that supports the use of pulmonary rehabilitation to decrease hospital admissions thereby reducing cost of care. Recent studies suggest that the significant benefits achieved through rehabilitation fade with time and that in order to improve activities of daily living; for example, average daily number of steps, programmes of longer duration are required.

The primary aim of this study is to identify objective sustained improved in activity levels using the SenseWear activity armband after a short-term pulmonary rehabilitation programme. Secondary aims are to determine antibiotic and steroid use pre and post rehabilitation.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is characterised by airflow limitation and by both systemic and airway inflammation. Together these features lead to decreased physical activity which in turn worsens the patient's dyspnoea. In patients with COPD, physical activity levels are low compared to healthy controls and indeed lower than in patients with other chronic conditions such as arthritis and diabetes. For patients with COPD, decreased physical activity and breathlessness are significant predictors of mortality and morbidity. By reversing deconditioning pulmonary rehabilitation using supervised and home exercise programs leads to increased exercise capacity and health quality of life scores. In order for the benefits of pulmonary rehabilitation to be sustained in the long-term it is essential that there is a change in the patient's physical activity in their home life. While practice guidelines recommend that there is transference of exercise to the home setting it is unknown if this happens in reality. Addressing whether there is an increase in physical activity at home after pulmonary rehabilitation is the focus of this study.

Physical activity can be measured in a number of ways, including direct observation, patient diaries and questionnaires, but one of the most successful are the performance based motion sensors such as pedometers and accelerometers. One such performance based motion sensor is the SenseWear accelerometer. The SenseWear has previously been used in patients with COPD, has been shown to be a reliable measure of physical activity performed in this population, other than those using rolators and it is objectively more accurate than questionnaires and diaries. The hypothesis of this study was that pulmonary rehabilitation leads to a sustained improvement in physical activity in patients with COPD. Physical activity was measured by the daily averaged activity recorded with a SenseWear armband at several time points in the year after a course of pulmonary rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of COPD based on the GOLD staging of the disease
* Referred to pulmonary rehabilitation by a respiratory consultant or member of the COPD Team
* Modified Medical Research Council Score of 3 or above
* Ability to mobilize independently
* Motivated to exercise independently

Exclusion Criteria:

* No evidence of COPD on spirometry
* Acute exacerbation within the last 4-6 weeks
* Evidence of ischemic heart disease/acute changes on ECG
* Uncontrolled hypertension
* Insulin dependent diabetes mellitus
* Inability to exercise independently or musculoskeletal/neurological conditions which would prevent completion of the course
* Lung cancer previous attendance at pulmonary rehabilitation

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2007-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Sustained improvement in free-living activities, measured as the average daily METs | At the end of 1 year compared to baseline
  Using an accelerometer, which will be worn by patients for seven consecutive days at each time frame, daily average measurements of the number of steps per day, total energy expenditure and METs that will be broken down into sedentary, moderate and vigorous, plus sleep time and efficiency.

SECONDARY OUTCOMES:
Quality of Life | baseline will be compared to that at 1 year follow-up
  Two quality of life questionnaires will be utilized, 1) the St. Georges Disease Questionnaire; a disease specific questionnaire, 2)The generic EuroQol questionnaire
The Incremental Shuttle Walk Test | baseline will be compared to that at 1 year follow-up
  This is a validated field exercise test used to prescribe exercise intensity and determine functional capacity
The Modified Medical Research Council Scale | baseline will be compared to that at 1 year follow-up
  This questionnaire measures breathlessness on activity
Pulmonary Function Tests | baseline will be compared to that at 1 year follow-up
  Measurements of forced expiratory volume in 1 second, Forced Vital Capacity, Inspiratory Capacity and peak inspiratory muscle pressure will all be measured
Borg Score | baseline will be compared to that at 1 year follow-up
  A 10 point scale measurement of breathlessness

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Costello, Professor, Study Chair — Beaumont Hospital; Brenda M Deering, MSc Physio, Principal Investigator — Beaumont Hospital; Claire Egan, MSc Physio, Principal Investigator — Beaumont Hospital; Niamh M McCormack, MSc Nursing, Principal Investigator — Beaumont Hosptial
Locations (1):
- Beaumont Hospital, Beaumont, Dublin, Ireland